CLINICAL TRIAL: NCT02987608
Title: A Feasibility Trial of Power Up: A Smartphone App to Support Young People to Make Shared Decisions in Therapy
Brief Title: A Feasibility Trial of Power Up
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: Anna Freud National Centre for Children and Families (Other); MindTech Healthcare Technology Co-operative (Unknown); Common Room Consulting Ltd (Unknown); Create Marketing (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16/0087
Record Dates: First submitted 2016-10-12; First posted 2016-12-09 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-10

CONDITIONS: Emotional Difficulties

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Phase (No Power Up) (No Intervention): 60 young people will receive CAMHS treatment as usual. Measures of empowerment, activation, and symptoms will be completed by participants soon after their referral to the service. The same measures plus shared decision making questionnaires will be administered three months later.
- Intervention Phase (Power Up) (Experimental): 60 young people use Power Up alongside CAMHS treatment as usual. Measures of empowerment, activation, and symptoms will be completed by participants soon after their referral to the service. The same measures plus shared decision making questionnaires and a Power Up feedback form will be administered three months later.
  Interventions: Device: Power Up

INTERVENTIONS:
Device: Power Up — Smartphone phone app
  Arms: Intervention Phase (Power Up)

SUMMARY:
There is an increasing demand for digital tools to empower young people with mental health difficulties (NHS England, 2015). Digital information, advice and mood tracking tools are increasingly being used to support child mental health. Evidence suggests that young people want to be active participants in their care and involved in decisions about their treatment. However, there is a lack of digital shared decision making tools available to support young people in Child and Adolescent Mental Health Services (CAMHS). This study aims to develop Power Up, a smartphone app to empower young people in CAMHS to make their voice heard and to participate more in decisions around their care.

The project will involve two phases:

* Development Phase -Developing Power Up according to the views and ideas expressed by young people, their parents/ carers, and clinicians in Patient and Public Involvement (PPI) sessions. -Conducting interviews and focus groups with 10 young people in CAMHS, 10 parents/ carers and 10 clinicians to review the acceptability of the content and format of Power Up.
* Feasibility testing Phase -Conducting a feasibility trial with 120 young people with emotional difficulties, aged 11-19 years, from three London CAMHS. 60 young people will receive treatment as usual and 60 will use Power Up alongside treatment as usual. Participant's ratings of empowerment, activation, and symptoms will be measured soon after their referral to the service. The same measures plus shared decision making questionnaires will be administered three months later.

The findings will inform the planning of a prospective cluster controlled trial. More broadly this trial will contribute an understanding of the feasibility and acceptability of developing and implementing a shared decision making app into CAMHS.

ELIGIBILITY:
Inclusion Criteria:

* Recently been referred to CAMHS (pre - first appointment)
* Presenting with emotional difficulties
* Clinician will have confirmed that the young person does not have any vulnerability which would make taking part in the study inappropriate to their context

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Shared Decision Making Questionnaire - 9 (SDM Q-9) | 3 months
  This will be completed by young people at time two (three months into therapy). The SDM Q-9 is a nine item patient reported shared decision making questionnaire.
CollaboRATE | 3 months
  This will be completed by young people at time two (three months into therapy). CollaboRATE is a three item patient reported shared decision making measure.
Experience of Service Questionnaire (ESQ) | 3 months
  Four items from this questionnaire will be completed by young people at time two (three months into therapy) as a proxy measure of shared decision making. The ESQ is a self-completion questionnaire that assesses children and young people's views of services with respect to accessibility, humanity of care, organisation of care and environment.
Dyadic OPTION scale | 3 months
  This will be completed by clinicians at time two (three months into therapy). The Dyadic OPTION scale is a 12- item instrument to measure the extent to which patients have been involved in shared decision making from the viewpoint of the clinician.

SECONDARY OUTCOMES:
Patient Activation Measure - Mental Health (PAM - MH) | 3 months
  The PAM - MH will be completed by young people at time one (beginning of therapy) and time two (three months into therapy). The PAM - MH is a patient reported tool for measuring engagement in mental healthcare.
Strengths and Difficulties questionnaire (SDQ) | 3 months
  The SDQ will be completed by young people at time one (beginning of therapy) and time two (three months into therapy). The SDQ is a self-report behavioural screening questionnaire for children and adolescents measuring symptoms and functioning.
Youth Efficacy / Empowerment Scale - Mental Health (YES - MH) | 3 months
  The YES -MH will be completed by young people at time one (beginning of therapy) and time two (three months into therapy). The YES - MH assesses youth perceptions of efficacy with respect to managing their own mental health condition ('Self'), managing their own services and supports ('Service'), and using their experience and knowledge to help peers and improve service systems ('System').
Client Receipt of Services Inventory (CSRI) - Children's Version. | 3 months
  The CSRI will be completed by parents at time one (beginning of therapy) and time two (three months into therapy). The CSRI provides information on service utilisation, as reported by the main carer of the child in the family.

OTHER OUTCOMES:
Did Not Attends (DNAs) | 3 months
  Number of young person DNAs will be reported by the clinician.
Number of sessions attended | 3 months
  The number of sessions attended by the young person will be reported by the clinician.
Type of therapy / intervention received | 3 months
  The type of therapy / intervention received by the young person will be reported by the clinician.

CONTACTS AND LOCATIONS:
Overall Officials: Miranda Wolpert, Professor, Principal Investigator — UCL & Anaa Freud National Centre for Children and Families
Locations (3):
- United Kingdom (3):
  - East London NHS Foundation Trust, London
  - North East London NHS Foundation Trust, London
  - The Tavistock and Portman NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chapman L, Edbrooke-Childs J, Martin K, Webber H, Craven MP, Hollis C, Deighton J, Law R, Fonagy P, Wolpert M. A Mobile Phone App to Support Young People in Making Shared Decisions in Therapy (Power Up): Study Protocol. JMIR Res Protoc. 2017 Oct 30;6(10):e206. doi: 10.2196/resprot.7694. PMID 29084708